CLINICAL TRIAL: NCT01247441
Title: Breast Cancer Registry - National University Health System, Singapore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR02/11/10
Record Dates: First submitted 2010-08-26; First posted 2010-11-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
Keywords: All breast cancer patients who were diagnosed or managed in NUH will be included into this registry
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Clinical data

SUMMARY:
The Breast Cancer Registry aims to collect clinical data of all breast cancer patients diagnosed and/or treated in the National University Hospital, with the goal of understanding risk factors, presenting symptoms, diagnosis, treatment, and outcome data of breast cancer in Singapore. This information will contribute to improving management of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- All breast cancer patients who were diagnosed or managed in NUH.

Exclusion Criteria:

- Non breast cancer patients.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Probability Sample
Dates: Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Dabakuyo TS, Bonnetain F, Roignot P, Poillot ML, Chaplain G, Altwegg T, Hedelin G, Arveux P. Population-based study of breast cancer survival in Cote d'Or (France): prognostic factors and relative survival. Ann Oncol. 2008 Feb;19(2):276-83. doi: 10.1093/annonc/mdm491. Epub 2007 Oct 24. PMID 17962200
- [Background] Park YH, Kim ST, Cho EY, Choi YL, Ok ON, Baek HJ, Lee JE, Nam SJ, Yang JH, Park W, Choi DH, Huh SJ, Ahn JS, Im YH. A risk stratification by hormonal receptors (ER, PgR) and HER-2 status in small (< or = 1 cm) invasive breast cancer: who might be possible candidates for adjuvant treatment? Breast Cancer Res Treat. 2010 Feb;119(3):653-61. doi: 10.1007/s10549-009-0665-x. PMID 19957028